CLINICAL TRIAL: NCT06774235
Title: Prevention of Secondary Infections by Interferon Gamma in ICU-acquired Sustained Immune-suppression: a Randomized Trial
Brief Title: Prevention of Secondary Infections by Interferon Gamma in ICU-acquired Sustained Immune-suppression
Acronym: PLATINIUM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 87RI24_0040 (PLATINIUM); 2024-516780-93-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-06; First posted 2025-01-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sustained Immunosuppression
Keywords: ICU; Immuno-restauration; Secondary infections; Prevention
MeSH Terms: conditions — Coinfection | interventions — Interferon-gamma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interferon-gamma (Experimental): Injections of Interferon gamma-1b are sub-cutaneous and preferably in the deltoid region left or right or on the anterior part of the thigh.
  5 injections between day 1 and day 9
  Interventions: Drug: Interferon Gamma 1-b
- Placebo (Placebo Comparator): The comparative treatment will be a placebo, consisting in 0.5 ml of 0.9% sodium chloride solution only (same volume for interferon gamma-1b)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon Gamma 1-b — injection of interferon gamma 1-b
  Arms: Interferon-gamma
Drug: Placebo — Injection of placebo in the same condition of experimental traitment
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to demonstrate the benefit of a standardized immunotherapy (Interferon gamma) on the incidence of secondary infections. . It will also learn about the safety of Interferon-gamma. The main questions it aims to answer are:

Does Interferon-gamma:

* reduces the Incidence of secondary infection episodes at three months
* reduces the ICU mortality and at Day 90
* reduces the ICU and hospital length of stay
* induces Biological immune restoration at Day 10
* has cost-consequence and cost-effectiveness

Researchers will compare Interferon-gamma to a placebo (a look-alike substance that contains no drug) to see if Interferon-gamma works to treat sustained immunosuppression .

Participants will:

* Take Interferon-Gamma or a placebo for a maximum of 5 times between day 1 and day 9
* be monitored evety day until their ICU discharge and at day 30, 60 and 90

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized in the ICU for at least 1 week
* Expected length of stay in the ICU greater than 10 days at screening
* At least 1 episode of multiple organ failure, defined as a SOFA ≥ 6 (excluding the respiratory component when related to a neurological failure), during the first 1 week of ICU hospitalization
* Immunosuppression defined as an mHLA-DR < 8000 Ab/c and a lymphopenia < 1000/mm3 within a 96 hours time window
* Patient or the legal representative giving consent must be able to understand the trial in its entirety
* Patient affiliated to the social security system
* For female participants of childbearing potential, agreement to use dual methods of contraception until Day 90
* For male participants with female partners of childbearing potential, agreement to use barrier method of contraception until Day 90.

Exclusion Criteria:

* Uncontrolled secondary infections ongoing at the time of screening
* Participation in another research clinical trial within 30 days
* Chemotherapy / radiation therapy within the last 6 weeks
* Apache II ≥ 30 at screening
* History of autoimmune disease
* Organ or bone marrow transplant
* History of hematologic malignancy
* History of hepatitis C
* HIV stage C within the last 12 months
* Patients under legal protection
* History of or ongoing tuberculosis
* Chronic hepatitis B
* Patients receiving immunosuppressive medications including patient receiving a steroid dose greater than 1mg/kg/day of prednisone equivalent for more than 1 week and patient that have been on corticosteroid for more than 3 months
* Patient with thrombocytopenia below 50,000/mm3
* Patient with traumatic brain and spinal injury
* Pregnancy or breast feeding
* Subjects with a history hypersensitivity to interferon gamma or excipient (Mannitol, Sodium succinate dibasic hexahydrate, Succinic acid, polysorbate 20), known latex hypersensitivity or other interferon
* Hepatic cytolysis with AST/ALT > 5 times ULN (local laboratory)
* Suspected acute pancreatitis with lipase or amylase > 3 times ULN (local laboratory)
* Severe chronic renal failure (eGFR<10 ml/min/1.73m2 CKP-EPI method)
* Acute ECG abnormality such as myocardial infarction or any acute life-threatening ECG abnormalities (e.g: ventricular fibrillation, ventricular tachycardia…)
* Mental state rendering the person giving consent incapable of understanding the trial
* Patient deprived of liberty by judicial or administrative decision
* Patient being the investigator, or any member of the team or relative of the investigator directly involved in the trial, including assistant doctors, pharmacists, nurses, trial coordinators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-10-09 (Estimated); Study Completion 2028-10-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of secondary infection episodes | Day 90
  Number of episodes divided by the follow-up length, in days, validated by an independent adjudication committee based on the current definitions.

SECONDARY OUTCOMES:
Cause of mortality of participant | Day 90
  All-cause ICU mortality and at Day 90
Length of stay in the ICU and in the hospital | Day 90
  Number of days spent in the ICU and in the hospital at Day 90
Antibiotic consumption | Day 90
  Name of antibiotics taken at Day 90
Biological immune restoration | Day 10
  Percentage of biological immune restoration (defined as an HLA-DR > 13 500 Ab/c [Antibodies bound per cell] and an absolute lymphocyte count > 1200 mm3) at Day 10
Healthcare costs | Day 90
  Healthcare costs at Day 90, cost per secondary infection avoided and cost per additional survivor, isolation requirement and antibiotic resistance
Rate of serious adverse reactions and suspected unexpected serious adverse reaction (SUSAR) | Day 90
  Rate of serious adverse reactions and suspected unexpected serious adverse reaction (SUSAR) at D90 according to sponsor causality assessment
Antifungal consumption | Day 90
  Name of antifungals taken at Day 90
Antifungal consumption | Day 90
  Dosage of antifungals taken at Day 90
Antifungal consumption | Day 90
  Duration of antifungals taken at Day 90
Antibiotic consumption | Day 90
  Dosage of antibiotics taken at Day 90
Antibiotic consumption | Day 90
  Duration of antibiotics taken at Day 90

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - Angers university hospial, Angers
  - Argenteuil hospital, Argenteuil
  - Franche-comté north Hospital, Belfort
  - Brive Hospital, Brive-la-Gaillarde
  - Chalon sur saone Hospital, Chalon-sur-Saône
  - Dijon University Hospital, Dijon
  - APHP - Raymond Poincaré, Garches
  - Versailles Hospital, Le Chesnay
  - Le mans Hospital, Le Mans
  - CH de Lens, Lens
  - Limoges University Hospital, Limoges
  - Lyon Civils Hospices, Lyon
  - APHM, Marseille
  - Melun Hospital, Melun
  - Nancy University Hospital, Nancy
  - Nantes University Hospital, Nantes
  - Orléans Hospital, Orléans
  - APHP - Laroiboisière, Paris
  - Aphp - Hegp, Paris
  - APHP - Cochin, Paris
  - Rennes University Hospital, Rennes
  - Strasbourg University Hospital, Strasbourg
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez Padilla AC, Daix T, Hotchkiss RS, Monneret G, Tadie JM, Jeannet R, Plateker O, Vaidie J, Durand-Zaleski I, Magne J, Giraudeau B, Francois B. Prevention of secondary infections by interferon-gamma in ICU-acquired sustained immune suppression in France: study protocol of the PLATINIUM randomised trial. BMJ Open. 2026 Jan 27;16(1):e106790. doi: 10.1136/bmjopen-2025-106790. PMID 41592843